CLINICAL TRIAL: NCT04740034
Title: A Multicenter, Phase 1, Open-label, Dose-escalation and Expansion Study of AMG 340, a Bispecific Antibody Targeting PSMA in Subjects With Metastatic Castrate-Resistant Prostate Carcinoma
Brief Title: A Study of AMG 340 in Subjects With Metastatic Castrate-Resistant Prostate Carcinoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor strategic decision
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TNB585.001; 20210249 (Other: Amgen)
Record Dates: First submitted 2021-02-01; First posted 2021-02-05 (Actual); Results first posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-05

CONDITIONS: Metastatic Castration-resistant Prostate Cancer
Keywords: Prostate specific membrane antigen; PSMA; Prostate cancer; Metastatic; Castrate-resistant
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation (Experimental): Sequential dose escalation cohorts are planned until maximum tolerated dose (MTD) is reached or recommended phase 2 dose (RP2D) is identified.
  Interventions: Drug: AMG 340
- Dose Expansion (Experimental): An expansion cohort in subjects with mCRPC will be enrolled after RP2D is established.
  Interventions: Drug: AMG 340

INTERVENTIONS:
Drug: AMG 340 — AMG 340 is a bispecific antibody targeting prostate-specific membrane antigen (PSMA) on tumor cells and CD3 on T-cells

SUMMARY:
This is a phase 1, open-label study evaluating the safety, clinical pharmacology and clinical activity of AMG 340, a PSMA x CD3 T-cell engaging bispecific antibody, in subjects with metastatic castrate-resistant prostate cancer (mCRPC) who have received 2 or more prior lines of therapy. The study consists of 2 parts, a monotherapy dose escalation (Arm A) and a monotherapy dose expansion (Arm B). Once the maximum tolerated dose (MTD) or recommended phase 2 dose (RP2D) is identified in Arm A, Arm B will be initiated to further characterize the safety, tolerability and pharmacokinetic (PK) profile of the MTD/RP2D dose of AMG 340 monotherapy in subjects with mCRPC.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed prostatic adenocarcinoma.
* History of metastatic disease.
* Chemically or surgically castrate.
* Subject has received at least 2 lines of systemic therapy approved for mCRPC, with disease progression on the most recent systemic therapy as defined in Prostate Cancer Working Group 3 (PCWG3) recommendations.
* Human immunodeficiency virus (HIV), hepatitis B virus (HBV), and/or hepatitis C virus (HCV)-infected subjects that have been cured or who are on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
* An Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 2.
* Subject must have adequate heart, liver, bone marrow and kidney function (e.g. estimated glomerular filtration rate [eGFR] ≥ 50 mL/min, aspartate aminotransferase [AST]/alanine aminotransferase [ALT] ≤ 3 x upper limit of normal [ULN], hemoglobin [Hgb] ≥ 9 g/dL (without blood transfusion within 7 days from screening assessment), platelets ≥ 100,000 / mm^3 (without platelet transfusion within 7 days from screening assessment), absolute neutrophil count [ANC] ≥ 1500 / mm^3).

Exclusion Criteria:

* Subject has been diagnosed with or treated for another malignancy within the past 2 years whose natural history or treatment may interfere with the safety or efficacy assessment of the investigational regimen.
* History of neuroendocrine differentiation in the subject's disease.
* Subject has a history of central nervous system (CNS) involvement by their mCRPC. Metastases stemming from bone are allowed.
* Subject has clinically significant CNS pathology.
* Subject requires chronic immunosuppressive therapy.
* Subject has a history of major cardiac abnormalities.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-04-29 (Actual); Primary Completion 2024-06-24 (Actual); Study Completion 2024-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (7):
- United States (7):
  - UCSF, San Francisco, California
  - Sarah Cannon Research Institute at HealthONE, Denver, Colorado
  - Florida Cancer Specialists, Sarasota, Florida
  - Tulane Cancer Center, New Orleans, Louisiana
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Thomas Jefferson University - Sidney Kimmel Cancer Center, Philadelphia, Pennsylvania
  - Tennessee Oncology, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with progressive metastatic castrate-resistant prostate carcinoma (mCRPC) participated in the study from April 2021 to June 2024, and were enrolled across 6 sites in the United States.
Pre-assignment Details: The study was designed to consist of two parts: a monotherapy dose escalation (Part A) and a monotherapy dose expansion (Part B). For strategic reasons, the study was terminated before enrollment into Part B could begin. Dose A is the lowest dose, Dose I is the highest dose.
Groups:
- Cohort 1: AMG 340 Dose A: Participants with progressive mCRPC received AMG 340 Dose A administered as an intravenous (IV) infusion every 3 week (Q3W) in 21-day cycles.
- Cohort 2: AMG 340 Dose B: Participants with progressive mCRPC received AMG 340 Dose B administered as an IV infusion Q3W in 21-day cycles.
- Cohort 3: AMG 340 Dose C: Participants with progressive mCRPC received AMG 340 Dose C administered as an IV infusion Q3W every 21-day cycle.
- Cohort 4: AMG 340 Dose D: Participants with progressive mCRPC received AMG 340 Dose D administered as an IV infusion Q3W in 21-day cycles.
- Cohort 5: AMG 340 Dose E: Participants with progressive mCRPC received AMG 340 Dose E administered as an IV infusion Q3W in 21-day cycles.
- Cohort 6a: AMG 340 Priming Dose (PmD) (High) and Then AMG 340 Dose E: Participants with progressive mCRPC received AMG 340 (high) PmD on Day 1 followed by AMG 340 Dose E on Day 8, both administered as IV infusions Q3W in 21-day cycles.
  Following protocol amendment 5 (07 Dec 2022), a second priming dose was added on Cycle 1 Day 5.
- Cohort 6b: AMG 340 PmD (Low) and Then AMG 340 Dose E: Participants with progressive mCRPC received AMG 340 PmD (low) on Day 1 followed by AMG 340 Dose E on Day 8, both administered as IV infusions Q3W in 21-day cycles.
  Following protocol amendment 5 (07 Dec 2022), a second priming dose was added on Cycle 1 Day 5.
- Cohort 7a: AMG 340 PmD (High) and Then AMG 340 Dose F: Participants with progressive mCRPC received AMG 340 PmD (high) on Day 1 followed by AMG 340 Dose F on Day 8, both administered as IV infusions Q3W in 21-day cycles.
  Following protocol amendment 5 (07 Dec 2022), a second priming dose was added on Cycle 1 Day 5.
- Cohort 8a: AMG 340 PmD (High) and Then AMG 340 Dose G: Participants with progressive mCRPC received AMG 340 PmD (high) on Day 1 followed by AMG 340 Dose G on Day 8, both administered as IV infusions Q3W in 21-day cycles.
  Following protocol amendment 5 (07 Dec 2022), a second priming dose was added on Cycle 1 Day 5.
- Cohort 9: AMG 340 PmD (High) and Then AMG 340 Dose H: Participants with progressive mCRPC received AMG 340 PmD (high) on Day 1 followed by AMG 340 Dose H on Day 8, both administered as IV infusions Q3W in 21-day cycles.
  Following protocol amendment 5 (07 Dec 2022), a second priming dose was added on Cycle 1 Day 5.
- Cohort 10: AMG 340 PmD (High) and Then AMG 340 Dose H and Dose I: Participants with progressive mCRPC received AMG 340 PmD (high) on Day 1 followed by AMG 340 Dose H and Dose I on Day 8, all doses were administered as IV infusions Q3W in 21-day cycles.
  Following protocol amendment 5 (07 Dec 2022), a second priming dose was added on Cycle 1 Day 5.
Period: Overall Study
Arm/Group | Cohort 1: AMG 340 Dose A | Cohort 2: AMG 340 Dose B | Cohort 3: AMG 340 Dose C | Cohort 4: AMG 340 Dose D | Cohort 5: AMG 340 Dose E | Cohort 6a: AMG 340 Priming Dose (PmD) (High) and Then AMG 340 Dose E | Cohort 6b: AMG 340 PmD (Low) and Then AMG 340 Dose E | Cohort 7a: AMG 340 PmD (High) and Then AMG 340 Dose F | Cohort 8a: AMG 340 PmD (High) and Then AMG 340 Dose G | Cohort 9: AMG 340 PmD (High) and Then AMG 340 Dose H | Cohort 10: AMG 340 PmD (High) and Then AMG 340 Dose H and Dose I
Started | 1 | 1 | 3 | 5 | 6 | 6 | 3 | 5 | 3 | 7 | 2
Completed | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 1 | 3 | 4 | 6 | 6 | 3 | 5 | 3 | 7 | 2
Not completed — Death | 0 | 1 | 2 | 3 | 4 | 4 | 2 | 2 | 2 | 4 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Decision by sponsor | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Population: Safety analysis set (SAS): All participants who received at least 1 dose of AMG 340.
Groups:
- Cohort 1: Dose A: Participants with progressive mCRPC received Dose A of AMG 340 administered as an intravenous (IV) infusion every 3 week (Q3W).
- Cohort 2: Dose B: Participants with progressive mCRPC received Dose B of AMG 340 administered as an IV infusion Q3W.
- Cohort 3: Dose C: Participants with progressive mCRPC received Dose C of AMG 340 administered as an IV infusion Q3W.
- Cohort 4: Dose D: Participants with progressive mCRPC received Dose D of AMG 340 administered as an IV infusion Q3W.
- Cohort 5: Dose E: Participants with progressive mCRPC received Dose E of AMG 340 administered as an IV infusion Q3W.
- Cohort 6a: AMG 340 PmD (High) and Then AMG 340 Dose E: Participants with progressive mCRPC received AMG 340 PmD (high) on Day 1 followed by AMG 340 Dose E on Day 8, both administered as IV infusions Q3W.
  Following protocol amendment 5 (07 Dec 2022), a second priming dose was added on Cycle 1 Day 5.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Dose A | Cohort 2: Dose B | Cohort 3: Dose C | Cohort 4: Dose D | Cohort 5: Dose E | Cohort 6a: AMG 340 PmD (High) and Then AMG 340 Dose E | Cohort 6b: AMG 340 PmD (Low) and Then AMG 340 Dose E | Cohort 7a: AMG 340 PmD (High) and Then AMG 340 Dose F | Cohort 8a: AMG 340 PmD (High) and Then AMG 340 Dose G | Cohort 9: AMG 340 PmD (High) and Then AMG 340 Dose H | Cohort 10: AMG 340 PmD (High) and Then AMG 340 Dose H and Dose I | Total
Number analyzed (Participants) | 1 | 1 | 3 | 5 | 6 | 6 | 3 | 5 | 3 | 7 | 2 | 42
Age, Continuous [Mean (Standard Deviation); unit: Years] | 78.0 (NA) — Not estimable due to only one participant in the analysis. | 54.0 (NA) — Not estimable due to only one participant in the analysis. | 69.0 (1.7) | 67.6 (7.4) | 71.8 (9.2) | 59.2 (6.4) | 75.7 (9.0) | 70.8 (5.2) | 67.0 (2.6) | 69.9 (4.5) | 71.0 (12.7) | 68.5 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 1 | 1 | 3 | 5 | 6 | 6 | 3 | 5 | 3 | 7 | 2 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 1 | 3 | 5 | 6 | 6 | 3 | 4 | 3 | 7 | 2 | 41
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 3
  White | 1 | 1 | 3 | 5 | 5 | 5 | 3 | 5 | 2 | 6 | 2 | 38
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical study participant, regardless of a causal relationship with the study treatment. TEAEs included any event occurring after the participant received the study treatment. A treatment-related AE (TRAE) was defined as any TEAE flagged as possibly caused by AMG 340. Clinically significant changes in vital signs, electrocardiograms, and laboratory tests recorded after treatment administration were documented as TEAEs. Serious TEAEs (SAEs) were any untoward medical occurrences after the first dose, irrespective of a causal link to the study treatment, that led to death, were life-threatening, required hospitalization or its prolongation, caused significant disability, resulted in congenital anomalies, or were considered other medically important events.
Time Frame: From enrollment up to and including a maximum of 90 days after last dose of AMG 340; median (min, max) duration was 4.3 (0.5, 27.1) months
Population: SAS: All participants who received at least 1 dose of AMG 340.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Dose A | Cohort 2: Dose B | Cohort 3: Dose C | Cohort 4: Dose D | Cohort 5: Dose E | Cohort 6a: AMG 340 PmD (High) and Then AMG 340 Dose E | Cohort 6b: AMG 340 PmD (Low) and Then AMG 340 Dose E | Cohort 7a: AMG 340 PmD (High) and Then AMG 340 Dose F | Cohort 8a: AMG 340 PmD (High) and Then AMG 340 Dose G | Cohort 9: AMG 340 PmD (High) and Then AMG 340 Dose H | Cohort 10: AMG 340 PmD (High) and Then AMG 340 Dose H and Dose I
Number analyzed (Participants) | 1 | 1 | 3 | 5 | 6 | 6 | 3 | 5 | 3 | 7 | 2
Participants
  All TEAEs | 1 | 1 | 3 | 5 | 6 | 6 | 3 | 5 | 3 | 7 | 2
  All SAEs | 0 | 0 | 2 | 3 | 3 | 4 | 2 | 1 | 2 | 4 | 0
  All TRAEs | 0 | 0 | 3 | 5 | 6 | 6 | 3 | 5 | 3 | 7 | 2

2. Primary Outcome: Number of Participants Who Experienced Dose Limiting Toxicities (DLTs)
Description: A DLT was defined as a TEAE that was not unequivocally due to the participant's underlying malignancy or other extraneous cause, and appeared within 21 days from the first dose of AMG 340. AEs considered DLTs were:
  * Transient (≤72 hours) grade 3 or 4 electrolyte abnormalities, hyperglycemia, nausea/vomiting/diarrhea responsive to treatment.
  * Alopecia, vitiligo, and grade 3 fatigue lasting <10 days.
  * Grade 3 fever lasting ≤24 hours (outside CRS context).
  * Grade 3 lab abnormalities resolving within 72 hours (or within 7 days for certain enzymes like ALT, GGT, ALP, and lipase).
  * Grade 3 CRS or TLS unresolved to ≤ grade 1 within 72 hours or any grade 4 CRS/TLS.
  * Prolonged grade 4 neutropenia (>5 days) or febrile neutropenia.
  * Grade 3 thrombocytopenia with bleeding or any grade 4 thrombocytopenia.
  * Grade 4 anemia.
  * Grade 5 adverse events.
  * Lymphopenia is not considered a DLT.
Time Frame: Up to approximately Day 21
Population: DLT evaluable analysis set: All participants who were evaluable for DLTs. A participants was considered DLT evaluable if the participant completed at least the first full treatment cycle or experienced a DLT during the first treatment cycle.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 6b: AMG 340 PmD (Low) and Then AMG 340 Dose E: Participants with progressive mCRPC received AMG 340 high PmD (low) on Day 1 followed by AMG 340 Dose E on Day 8, both administered as IV infusions Q3W in 21-day cycles.
  Following protocol amendment 5 (07 Dec 2022), a second priming dose was added on Cycle 1 Day 5.
Arm/Group | Cohort 1: Dose A | Cohort 2: Dose B | Cohort 3: Dose C | Cohort 4: Dose D | Cohort 5: Dose E | Cohort 6a: AMG 340 PmD (High) and Then AMG 340 Dose E | Cohort 6b: AMG 340 PmD (Low) and Then AMG 340 Dose E | Cohort 7a: AMG 340 PmD (High) and Then AMG 340 Dose F | Cohort 8a: AMG 340 PmD (High) and Then AMG 340 Dose G | Cohort 9: AMG 340 PmD (High) and Then AMG 340 Dose H | Cohort 10: AMG 340 PmD (High) and Then AMG 340 Dose H and Dose I
Number analyzed (Participants) | 1 | 1 | 2 | 5 | 5 | 6 | 3 | 5 | 3 | 6 | 2
Participants | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1

3. Primary Outcome: Median Concentration of AMG 340
Description: Blood samples for pharmacokinetics (PK) analysis were collected at specific time points. PK parameters were estimated using standard non-compartmental approaches.
Time Frame: Cohorts 1-5: Days 1 (pre-dose to 6 hours post-dose), 2, 3, 8, and 10; Cohorts 6-10: Days 1 (pre-dose to 6 hours post-dose), 2, 3, 5 (pre-dose to 6 hours post-dose), 6, 7, 8 (pre-dose to 6 hours post-dose), 9, 10
Population: PK analysis set: Included all participants who received at least 1 dose of AMG 340 and had at least 1 PK sample drawn post dose. Summary statistics are presented per dose level as pre-specified in SAP Section 9.7.
Measure: Median (Full Range); unit: µg/mL
Groups:
- Cohort 6: AMG 340 PmD (Low) and (High), and Then AMG 340 Dose E: Participants with progressive mCRPC received AMG 340 PmD (low) and (high) on Day 1 followed by AMG 340 Dose E on Day 8, both administered as IV infusions Q3W.
  Following protocol amendment 5 (07 Dec 2022), a second priming dose was added on Cycle 1 Day 5.
Arm/Group | Cohort 1: Dose A | Cohort 2: Dose B | Cohort 3: Dose C | Cohort 4: Dose D | Cohort 5: Dose E | Cohort 6: AMG 340 PmD (Low) and (High), and Then AMG 340 Dose E | Cohort 7a: AMG 340 PmD (High) and Then AMG 340 Dose F | Cohort 8a: AMG 340 PmD (High) and Then AMG 340 Dose G | Cohort 9: AMG 340 PmD (High) and Then AMG 340 Dose H | Cohort 10: AMG 340 PmD (High) and Then AMG 340 Dose H and Dose I
Number analyzed (Participants) | 1 | 1 | 3 | 5 | 6 | 9 | 5 | 3 | 3 | 2
µg/mL | 0.352 [0.352 to 0.352] | 0.818 [0.818 to 0.818] | 2.445 [0.233 to 4.71] | 6.78 [0.661 to 16.2] | 17.8 [0.116 to 54.5] | 19.25 [0 to 52.3] | 54.4 [3.61 to 129] | 68.0 [17.1 to 149] | 75.2 [2.64 to 201] | 201 [79.1 to 397]

4. Secondary Outcome: Percentage of Participants Who Achieved an Objective Response (OR) Per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
Description: OR was defined as a partial response (PR) or complete response (CR) per RECIST 1.1, confirmed by a repeat assessment at least 4 weeks later. Participants who did not experience a confirmed PR/CR or did not have any follow-up tumor assessments were regarded as non-responders.
Time Frame: Up to approximately 24 months
Population: RECIST 1.1 Evaluable Analysis Set: All participants who have received at least 1 dose of AMG 340, had measurable disease per RECIST 1.1 at baseline, and had the opportunity to be followed for at least 6 weeks from start of AMG 340 treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Cohort 7a: AMG 340 PmD A and Then AMG 340 Dose F: Participants with progressive mCRPC received AMG 340 PmD A on Day 1 followed by AMG 340 Dose F on Day 8, both administered as IV infusions Q3W in 21-day cycles.
  Following protocol amendment 5 (07 Dec 2022), a second priming dose was added on Cycle 1 Day 5.
Arm/Group | Cohort 1: Dose A | Cohort 2: Dose B | Cohort 3: Dose C | Cohort 4: Dose D | Cohort 5: Dose E | Cohort 6a: AMG 340 PmD (High) and Then AMG 340 Dose E | Cohort 6b: AMG 340 PmD (Low) and Then AMG 340 Dose E | Cohort 7a: AMG 340 PmD A and Then AMG 340 Dose F | Cohort 8a: AMG 340 PmD (High) and Then AMG 340 Dose G | Cohort 9: AMG 340 PmD (High) and Then AMG 340 Dose H | Cohort 10: AMG 340 PmD (High) and Then AMG 340 Dose H and Dose I
Number analyzed (Participants) | 0 | 0 | 3 | 2 | 4 | 4 | 2 | 3 | 2 | 5 | 2
Percentage of Participants |  |  | 0 [0.0 to 70.76] | 0 [0.0 to 84.19] | 0 [0.0 to 60.24] | 0 [0.0 to 60.24] | 0 [0.0 to 84.19] | 0 [0.0 to 70.76] | 0 [0.0 to 84.19] | 0 [0.0 to 52.18] | 0 [0.0 to 84.19]

5. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of study Day 1 until death due to any cause.
Time Frame: Up to approximately 24 months
Population: SAS: All participants who received at least 1 dose of AMG 340.
Measure: Median (Full Range); unit: Months
Arm/Group | Cohort 1: Dose A | Cohort 2: Dose B | Cohort 3: Dose C | Cohort 4: Dose D | Cohort 5: Dose E | Cohort 6a: AMG 340 PmD (High) and Then AMG 340 Dose E | Cohort 6b: AMG 340 PmD (Low) and Then AMG 340 Dose E | Cohort 7a: AMG 340 PmD (High) and Then AMG 340 Dose F | Cohort 8a: AMG 340 PmD (High) and Then AMG 340 Dose G | Cohort 9: AMG 340 PmD (High) and Then AMG 340 Dose H | Cohort 10: AMG 340 PmD (High) and Then AMG 340 Dose H and Dose I
Number analyzed (Participants) | 1 | 1 | 3 | 5 | 6 | 6 | 3 | 5 | 3 | 7 | 2
Months | 9.2 [9.2 to 9.2] | 13.4 [13.4 to 13.4] | 10.22 [4.8 to 12.2] | 11.56 [3.4 to 20.3] | 5.59 [1.6 to 19.2] | 8.15 [3.1 to 19.3] | 5.45 [4.2 to 25.7] | NA [3.0 to 28.2] — Median could not be calculated as there was an insufficient number of participants with events. | 6.97 [1.5 to 27.1] | 7.56 [0.5 to 15.4] | NA [8.5 to 10.6] — Median could not be calculated as there was an insufficient number of participants with events.

6. Secondary Outcome: Prostate Specific Antigen (PSA) Progression Free Survival (PFS)
Description: PSA PFS was defined as the interval from study day 1 to the earlier of a PSA progression or death from any cause; otherwise, PSA PFS was censored on the date of the last PSA measurement. If a participant had no baseline or post-baseline PSA measurement and a vital status of alive or unknown, PSA PFS was censored at study day 1.
Time Frame: Up to approximately 24 months
Population: SAS: All participants who received at least 1 dose of AMG 340.
Measure: Median (Full Range); unit: Months
Arm/Group | Cohort 1: Dose A | Cohort 2: Dose B | Cohort 3: Dose C | Cohort 4: Dose D | Cohort 5: Dose E | Cohort 6a: AMG 340 PmD (High) and Then AMG 340 Dose E | Cohort 6b: AMG 340 PmD (Low) and Then AMG 340 Dose E | Cohort 7a: AMG 340 PmD (High) and Then AMG 340 Dose F | Cohort 8a: AMG 340 PmD (High) and Then AMG 340 Dose G | Cohort 9: AMG 340 PmD (High) and Then AMG 340 Dose H | Cohort 10: AMG 340 PmD (High) and Then AMG 340 Dose H and Dose I
Number analyzed (Participants) | 1 | 1 | 3 | 5 | 6 | 6 | 3 | 5 | 3 | 7 | 2
Months | 1.4 [1.4 to 1.4] | 2.1 [2.1 to 2.1] | 4.83 [3.4 to 6.9] | 3.20 [2.1 to 6.2] | 2.89 [1.5 to 8.3] | 3.12 [1.9 to 8.1] | 2.8 [2.8 to 5.5] | 3.48 [0.0 to 3.8] | 6.97 [1.5 to 27.1] | 4.86 [0.0 to 9.4] | NA [1.4 to 1.9] — Median could not be calculated as there was an insufficient number of participants with events.

7. Secondary Outcome: Radiographic PFS (rPFS)
Description: rPFS was defined as the interval from study day 1 to radiographic progression or death from any cause, whichever occurred first, in the absence of subsequent anti-cancer therapy; otherwise, rPFS was censored at the last evaluable tumor assessment date prior to subsequent anti-cancer therapy.
  If a participant had no post-baseline radiographic tumor assessment and a vital status of alive or unknown, rPFS was censored at study day 1.
Time Frame: Up to approximately 24 months
Population: SAS: All participants who received at least 1 dose of AMG 340.
Measure: Median (Full Range); unit: Months
Arm/Group | Cohort 1: Dose A | Cohort 2: Dose B | Cohort 3: Dose C | Cohort 4: Dose D | Cohort 5: Dose E | Cohort 6a: AMG 340 PmD (High) and Then AMG 340 Dose E | Cohort 6b: AMG 340 PmD (Low) and Then AMG 340 Dose E | Cohort 7a: AMG 340 PmD (High) and Then AMG 340 Dose F | Cohort 8a: AMG 340 PmD (High) and Then AMG 340 Dose G | Cohort 9: AMG 340 PmD (High) and Then AMG 340 Dose H | Cohort 10: AMG 340 PmD (High) and Then AMG 340 Dose H and Dose I
Number analyzed (Participants) | 1 | 1 | 3 | 5 | 6 | 6 | 3 | 5 | 3 | 7 | 2
Months | NA [7.8 to 7.8] — Median could not be calculated as there was an insufficient number of participants with events. | 3.48 [3.48 to 3.48] | 5.32 [1.4 to 7.2] | 3.38 [1.2 to 3.4] | 1.56 [1.4 to 6.2] | 2.25 [0.9 to 9.4] | 4.27 [1.2 to 5.5] | 3.84 [1.4 to 7.5] | 1.31 [1.2 to 11.7] | 2.35 [0.00 to 13.6] | NA [1.9 to 3.9] — Median could not be calculated as there was an insufficient number of participants with events.

8. Secondary Outcome: Percentage of Participants With rPFS at 6 Months
Description: as for outcome 7
Time Frame: 6 months
Population: SAS: All participants who received at least 1 dose of AMG 340.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: Dose A | Cohort 2: Dose B | Cohort 3: Dose C | Cohort 4: Dose D | Cohort 5: Dose E | Cohort 6a: AMG 340 PmD (High) and Then AMG 340 Dose E | Cohort 6b: AMG 340 PmD (Low) and Then AMG 340 Dose E | Cohort 7a: AMG 340 PmD (High) and Then AMG 340 Dose F | Cohort 8a: AMG 340 PmD (High) and Then AMG 340 Dose G | Cohort 9: AMG 340 PmD (High) and Then AMG 340 Dose H | Cohort 10: AMG 340 PmD (High) and Then AMG 340 Dose H and Dose I
Number analyzed (Participants) | 1 | 1 | 3 | 5 | 6 | 6 | 3 | 5 | 3 | 7 | 2
Percentage of participants | 100.0 [NA to NA] — 95% Confidence interval (CI) not estimable due to the low number of participants in the analysis population. | 0.0 [NA to NA] — 95% CI not estimable due to the low number of participants in the analysis population. | 33.3 [0.9 to 77.4] | 0.0 [NA to NA] — 95% CI could not be calculated as there was an insufficient number of participants with events. | 33.3 [4.6 to 67.6] | 16.7 [0.8 to 51.7] | 0.0 [NA to NA] — 95% CI not estimable due to the low number of participants in the analysis population. | 33.3 [0.9 to 77.4] | 33.3 [0.9 to 77.4] | 16.7 [0.8 to 51.7] | NA [NA to NA] — Median and 95% CI not estimable due to the low number of participants in the analysis population.

9. Secondary Outcome: Percentage of Participants With a 30% Reduction From Baseline in PSA (PSA30)
Description: PSA 30 was defined as a ≥ 30% reduction from the baseline PSA. This PSA response had to be confirmed by a second consecutive value obtained at least three weeks later.
Time Frame: Up to approximately 24 months
Population: The PSA response evaluable analysis set was defined as all participants who received at least one dose of AMG 340, had a measurable (i.e., > 0) PSA at baseline, and had the opportunity to be followed for at least nine weeks from the start of AMG 340 treatment.
  Participants who stopped disease assessments prior to nine weeks were included in this analysis set if the data snapshot date was at least nine weeks after their first study dose date.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort 1: Dose A | Cohort 2: Dose B | Cohort 3: Dose C | Cohort 4: Dose D | Cohort 5: Dose E | Cohort 6a: AMG 340 PmD (High) and Then AMG 340 Dose E | Cohort 6b: AMG 340 PmD (Low) and Then AMG 340 Dose E | Cohort 7a: AMG 340 PmD (High) and Then AMG 340 Dose F | Cohort 8a: AMG 340 PmD (High) and Then AMG 340 Dose G | Cohort 9: AMG 340 PmD (High) and Then AMG 340 Dose H | Cohort 10: AMG 340 PmD (High) and Then AMG 340 Dose H and Dose I
Number analyzed (Participants) | 1 | 1 | 3 | 5 | 6 | 6 | 3 | 5 | 3 | 7 | 2
Percentage of Participants | 0.0 [0.00 to 97.50] | 100.0 [2.5 to 100.00] | 33.3 [0.84 to 90.57] | 20.0 [0.51 to 71.64] | 0.0 [0.00 to 45.93] | 16.7 [0.42 to 64.12] | 0.0 [0.00 to 70.76] | 20.0 [0.51 to 71.64] | 33.3 [0.84 to 90.57] | 0.0 [0.00 to 40.96] | 0.0 [0.00 to 84.19]

10. Secondary Outcome: Percentage of Participants With a 50% Reduction From Baseline in PSA (PSA50)
Description: PSA 50 was defined as a ≥ 50% reduction from the baseline PSA. This PSA response had to be confirmed by a second consecutive value obtained at least three weeks later.
Time Frame: Up to approximately 24 months
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort 1: Dose A | Cohort 2: Dose B | Cohort 3: Dose C | Cohort 4: Dose D | Cohort 5: Dose E | Cohort 6a: AMG 340 PmD (High) and Then AMG 340 Dose E | Cohort 6b: AMG 340 PmD (Low) and Then AMG 340 Dose E | Cohort 7a: AMG 340 PmD (High) and Then AMG 340 Dose F | Cohort 8a: AMG 340 PmD (High) and Then AMG 340 Dose G | Cohort 9: AMG 340 PmD (High) and Then AMG 340 Dose H | Cohort 10: AMG 340 PmD (High) and Then AMG 340 Dose H and Dose I
Number analyzed (Participants) | 1 | 1 | 3 | 5 | 6 | 6 | 3 | 5 | 3 | 7 | 2
Percentage of Participants | 0.0 [0.00 to 97.50] | 100.0 [2.5 to 100.0] | 33.3 [0.84 to 90.57] | 20.0 [0.51 to 71.64] | 0.0 [0.00 to 45.93] | 16.7 [0.42 to 64.12] | 0.0 [0.00 to 70.76] | 0.0 [0.00 to 52.18] | 0.0 [0.00 to 70.76] | 0.0 [0.00 to 40.96] | 0.0 [0.00 to 84.19]

11. Secondary Outcome: Percentage of Participants With a 70% Reduction From Baseline in PSA (PSA70)
Description: PSA 70 was defined as a ≥ 70% reduction from the baseline PSA. This PSA response had to be confirmed by a second consecutive value obtained at least three weeks later.
Time Frame: Up to approximately 24 months
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort 1: Dose A | Cohort 2: Dose B | Cohort 3: Dose C | Cohort 4: Dose D | Cohort 5: Dose E | Cohort 6a: AMG 340 PmD (High) and Then AMG 340 Dose E | Cohort 6b: AMG 340 PmD (Low) and Then AMG 340 Dose E | Cohort 7a: AMG 340 PmD (High) and Then AMG 340 Dose F | Cohort 8a: AMG 340 PmD (High) and Then AMG 340 Dose G | Cohort 9: AMG 340 PmD (High) and Then AMG 340 Dose H | Cohort 10: AMG 340 PmD (High) and Then AMG 340 Dose H and Dose I
Number analyzed (Participants) | 1 | 1 | 3 | 5 | 6 | 6 | 3 | 5 | 3 | 7 | 2
Percentage of Participants | 0.0 [0.00 to 97.50] | 0.0 [0.0 to 97.50] | 0.0 [0.0 to 70.76] | 0.0 [0.0 to 52.18] | 0.0 [0.00 to 45.93] | 0.0 [0.0 to 45.93] | 0.0 [0.00 to 70.76] | 0.0 [0.00 to 52.18] | 0.0 [0.00 to 70.76] | 0.0 [0.00 to 40.96] | 0 [0.00 to 84.19]

12. Secondary Outcome: Percentage of Participants With a 90% Reduction From Baseline in PSA (PSA90)
Description: PSA 90 was defined as a ≥ 90% reduction from the baseline PSA. This PSA response had to be confirmed by a second consecutive value obtained at least three weeks later.
Time Frame: Up to approximately 24 months
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort 1: Dose A | Cohort 2: Dose B | Cohort 3: Dose C | Cohort 4: Dose D | Cohort 5: Dose E | Cohort 6a: AMG 340 PmD (High) and Then AMG 340 Dose E | Cohort 6b: AMG 340 PmD (Low) and Then AMG 340 Dose E | Cohort 7a: AMG 340 PmD (High) and Then AMG 340 Dose F | Cohort 8a: AMG 340 PmD (High) and Then AMG 340 Dose G | Cohort 9: AMG 340 PmD (High) and Then AMG 340 Dose H | Cohort 10: AMG 340 PmD (High) and Then AMG 340 Dose H and Dose I
Number analyzed (Participants) | 1 | 1 | 3 | 5 | 6 | 6 | 3 | 5 | 3 | 7 | 2
Percentage of Participants | 0.0 [0.00 to 97.50] | 0.0 [0.00 to 97.50] | 0.0 [0.00 to 70.76] | 0.0 [0.00 to 52.18] | 0.0 [0.00 to 45.93] | 0.0 [0.00 to 45.93] | 0.0 [0.00 to 70.76] | 0.0 [0.00 to 52.18] | 0.0 [0.00 to 70.76] | 0.0 [0.00 to 40.96] | 0.0 [0.00 to 84.19]

13. Secondary Outcome: Duration of Response (DOR) Per RECIST 1.1
Description: DOR was defined as the time from the date of an initial objective response per RECIST 1.1, which was subsequently confirmed, until soft-tissue progression per RECIST 1.1 or death, whichever occurred first in the absence of subsequent anti-cancer therapy. Participants who had not ended their response at the time of analysis had DOR censored at their last evaluable tumor assessment by CT/MRI scan prior to subsequent anti-cancer therapy. This endpoint only applied to participants with an objective response (CR or PR) per RECIST 1.1. No participants achieved CR or PR, therefore, no participants could be analyzed for this outcome measure.
Time Frame: Up to approximately 24 months
Population: RECIST 1.1 Evaluable Analysis Set: All participants who received at least one dose of AMG 340, had measurable disease per RECIST 1.1 at baseline, and had the opportunity to be followed for at least six weeks from the start of AMG 340 treatment. Participants who stopped disease assessments prior to six weeks were included in this analysis set if the data snapshot date was at least six weeks after their first study dose date.
Arm/Group | Cohort 1: Dose A | Cohort 2: Dose B | Cohort 3: Dose C | Cohort 4: Dose D | Cohort 5: Dose E | Cohort 6a: AMG 340 PmD (High) and Then AMG 340 Dose E | Cohort 6b: AMG 340 PmD (Low) and Then AMG 340 Dose E | Cohort 7a: AMG 340 PmD (High) and Then AMG 340 Dose F | Cohort 8a: AMG 340 PmD (High) and Then AMG 340 Dose G | Cohort 9: AMG 340 PmD (High) and Then AMG 340 Dose H | Cohort 10: AMG 340 PmD (High) and Then AMG 340 Dose H and Dose I
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

14. Secondary Outcome: Number of Participants With Symptomatic Skeletal Events (SSE)
Description: SSE was defined as time from study day 1 to the first symptomatic skeletal event, otherwise time to symptomatic skeletal event was censored at the last dose of AMG 340 or end of safety follow-up date, whichever was later.
Time Frame: Up to approximately 24 months
Population: SAS: All participants who received at least 1 dose of AMG 340.
Measure: Number; unit: Number of Participants
Arm/Group | Cohort 1: Dose A | Cohort 2: Dose B | Cohort 3: Dose C | Cohort 4: Dose D | Cohort 5: Dose E | Cohort 6a: AMG 340 PmD (High) and Then AMG 340 Dose E | Cohort 6b: AMG 340 PmD (Low) and Then AMG 340 Dose E | Cohort 7a: AMG 340 PmD (High) and Then AMG 340 Dose F | Cohort 8a: AMG 340 PmD (High) and Then AMG 340 Dose G | Cohort 9: AMG 340 PmD (High) and Then AMG 340 Dose H | Cohort 10: AMG 340 PmD (High) and Then AMG 340 Dose H and Dose I
Number analyzed (Participants) | 1 | 1 | 3 | 5 | 6 | 6 | 3 | 5 | 3 | 7 | 2
Number of Participants | 0 | 0 | 1 | 1 | 2 | 2 | 0 | 1 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Death: From enrollment through end of study; median (min, max) time on study was 7.4 (0.5, 28.2) months. TEAE: From enrollment up to and including a maximum of 90 days after last dose of AMG 340; median (min, max) duration was 4.3 (0.5, 27.1) months.
Description: Serious adverse events and other adverse events are reported for all participants who received at least one dose of study drug. All-cause mortality is reported for all participants enrolled in the study.
Groups:
- Cohort 1: Dose A: Participants with progressive mCRPC received Dose A of AMG 340 administered as an IV infusion Q3W.
Arm/Group | Cohort 1: Dose A | Cohort 2: Dose B | Cohort 3: Dose C | Cohort 4: Dose D | Cohort 5: Dose E | Cohort 6a: AMG 340 PmD (High) and Then AMG 340 Dose E | Cohort 6b: AMG 340 PmD (Low) and Then AMG 340 Dose E | Cohort 7a: AMG 340 PmD (High) and Then AMG 340 Dose F | Cohort 8a: AMG 340 PmD (High) and Then AMG 340 Dose G | Cohort 9: AMG 340 PmD (High) and Then AMG 340 Dose H | Cohort 10: AMG 340 PmD (High) and Then AMG 340 Dose H and Dose I
All-Cause Mortality (participants affected / at risk) | 0/1 | 1/1 | 2/3 | 3/5 | 4/6 | 4/6 | 2/3 | 2/5 | 2/3 | 4/7 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 2/3 | 3/5 | 3/6 | 4/6 | 2/3 | 1/5 | 2/3 | 4/7 | 0/2
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 3/3 | 5/5 | 6/6 | 6/6 | 3/3 | 5/5 | 3/3 | 7/7 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Dose A (N=1) | Cohort 2: Dose B (N=1) | Cohort 3: Dose C (N=3) | Cohort 4: Dose D (N=5) | Cohort 5: Dose E (N=6) | Cohort 6a: AMG 340 PmD (High) and Then AMG 340 Dose E (N=6) | Cohort 6b: AMG 340 PmD (Low) and Then AMG 340 Dose E (N=3) | Cohort 7a: AMG 340 PmD (High) and Then AMG 340 Dose F (N=5) | Cohort 8a: AMG 340 PmD (High) and Then AMG 340 Dose G (N=3) | Cohort 9: AMG 340 PmD (High) and Then AMG 340 Dose H (N=7) | Cohort 10: AMG 340 PmD (High) and Then AMG 340 Dose H and Dose I (N=2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 3 | 0
Brain abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Dose A (N=1) | Cohort 2: Dose B (N=1) | Cohort 3: Dose C (N=3) | Cohort 4: Dose D (N=5) | Cohort 5: Dose E (N=6) | Cohort 6a: AMG 340 PmD (High) and Then AMG 340 Dose E (N=6) | Cohort 6b: AMG 340 PmD (Low) and Then AMG 340 Dose E (N=3) | Cohort 7a: AMG 340 PmD (High) and Then AMG 340 Dose F (N=5) | Cohort 8a: AMG 340 PmD (High) and Then AMG 340 Dose G (N=3) | Cohort 9: AMG 340 PmD (High) and Then AMG 340 Dose H (N=7) | Cohort 10: AMG 340 PmD (High) and Then AMG 340 Dose H and Dose I (N=2)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 1 | 2 | 2 | 1 | 1 | 0 | 3 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 2 | 1 | 2 | 3 | 2 | 1 | 2 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ear congestion (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 2 | 1 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 2 | 4 | 3 | 0 | 1 | 3 | 0 | 2 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 2 | 1 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 4 | 4 | 2 | 1 | 4 | 2 | 2 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 3 | 4 | 3 | 1 | 3 | 1 | 3 | 2
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chills (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 1
Fatigue (General disorders) | 1 | 0 | 2 | 2 | 2 | 0 | 1 | 4 | 1 | 5 | 1
Influenza like illness (General disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 1 | 3 | 0 | 2 | 0 | 1 | 1
Liver disorder (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 2 | 4 | 1 | 2 | 2 | 3 | 4 | 2
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Impetigo (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 3 | 4 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 2 | 3 | 4 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 3 | 2 | 0 | 1 | 0 | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 2 | 3 | 2 | 2 | 0 | 3 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3 | 1 | 3 | 1 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 2 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 1 | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Bell's palsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1 | 3 | 3 | 0 | 2 | 1 | 1 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 2 | 1 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Taste disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Depression (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Genital pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 1 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 2 | 1 | 1 | 2
Ex-tobacco user (Social circumstances) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 2 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2022-12-07): https://cdn.clinicaltrials.gov/large-docs/34/NCT04740034/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-31): https://cdn.clinicaltrials.gov/large-docs/34/NCT04740034/SAP_001.pdf